CLINICAL TRIAL: NCT05379751
Title: Tentacle Shaped Mesh for Fixation Free Spigelian Hernia Repair
Brief Title: Surgical Repair of Spigelian Hernia in a Cohort of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Giuseppe Amato, Consultant Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spigelian hernia treatment
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Spigelian Hernia

STUDY DESIGN:
Intervention Model Description: A cohort of 54 patients diagnosed with Spigelian hernia who underwent open surgical repair with the tentacle shaped implant (Freedom Octomesh VHR XS produced by Insightra Medical Inc. - USA) forms the body of this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients diagnosed with Spigelian hernia who underwent prosthetic repair with the tentacle mesh (Experimental): Patients diagnosed with Spigelian hernia who underwent prosthetic repair with the tentacle mesh Freedom Octomesh VHR XS
  Interventions: Procedure: Fixation free Spigelian hernia repair with tentacle mesh

INTERVENTIONS:
Procedure: Fixation free Spigelian hernia repair with tentacle mesh — Spigelian hernias are repaired through the fixation free placement of a tentacle mesh in preperitoneal sublay thanks the friction exerted by the tentacle straps delivered by a proprietary needle passer crossing trouh the abdominal wall from the preperitoneal space until the subutaneous layer. This procedural approach should also grant a broad overlap of the implant over the hernial defect

SUMMARY:
Repair of Spigelian hernias with a tentacle shaped implant and highlighting the results of the procedure

DETAILED DESCRIPTION:
The surgical treatment of Spigelian hernias is mainly carried out with prosthetic meshes made of biocompatible material. In prosthetic repair of abdominal protrusions, mesh fixation and overlap of the mesh are source of complications. To avoid these problems, for a fixation free repair of Spigelian hernias has been developed a tentacle shaped implant, that should also assure a broader defect overlap. This study should highlight in a cohort of patients the long-term results of fixation free repair of Spigelian hernias carried out with tentacle mesh.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Spigelian hernia

Exclusion Criteria:

* Patients not having Spigelian hernia,

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Fixation free prosthetic repair of Spigelian hernias with tentacle mesh | Intraoperative
  Feasibility of fixation free placement of tentacle mesh in Spigelian hernia repair
Granting a broad implant overlap in prosthetic repair of Spigelian hernias with tentacle mesh | between 6 and 84 months postop
  Granting a broad overlap over the hernial defect after placement in preperitoneal sublay of tentacle mesh in Spigelian hernia repair with tentacle mesh to reduce risks of recurrence in the long term postop.

SECONDARY OUTCOMES:
Intra-operative features | intraoperatively
  reduction of the operative time length
Postoperative features 1 | between 6 and 84 months postop
  Postoperative pain assessment with VAS scoring system
Postoperative features 2 | between 6 and 84 months postop
  Assessment of postoperative complications

IPD SHARING:
Plan to Share IPD: No